CLINICAL TRIAL: NCT01580891
Title: Randomized, Double-Blind, Placebo-Controlled, Multiple-Site, Parallel Design Study to Evaluate the Clinical Equivalence of Two Naftifine HCl 1% Creams in Patients With Interdigital Tinea Pedis.
Brief Title: Evaluate the Clinical Equivalence of Two Naftifine HCl 1% Creams in Patients With Interdigital Tinea Pedis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTFC 1105.0
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Tinea Pedis
Keywords: Naftifine HCl Cream 1%; Naftin® (Naftifine HCl) Cream 1%; Tinea Pedis; Efficacy and safety
MeSH Terms: conditions — Tinea Pedis | interventions — naftifine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Naftifine HCl Cream 1% (Experimental): Naftifine HCl Cream 1% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Naftifine HCl Cream 1%
- Naftin® (Naftifine HCl) Cream 1% (Active Comparator): Naftin® (Naftifine HCl) Cream 1% (Merz Pharmaceuticals)
  Interventions: Drug: Naftin® (Naftifine HCl) Cream 1%
- Placebo topical cream (Placebo Comparator): Placebo topical cream (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Placebo topical cream

INTERVENTIONS:
Drug: Naftifine HCl Cream 1% — Naftifine HCl Cream 1% applied topically once a day for 28 days.
  Arms: Naftifine HCl Cream 1%
Drug: Naftin® (Naftifine HCl) Cream 1% — Naftin® (Naftifine HCl) Cream 1% applied topically once a day for 28 days.
  Arms: Naftin® (Naftifine HCl) Cream 1%
Drug: Placebo topical cream — Placebo topical cream applied topically once a day for 28 days.
  Arms: Placebo topical cream

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of the test formulation of Naftifine HCl Cream 1% (Taro Pharmaceuticals Inc.) as compared to the already marketed formulation Naftin® (Naftifine HCl) 1% Cream (Merz Pharmaceuticals) and placebo in patients with tinea pedis and to show the superiority of the active treatments over placebo when dosed once a day for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females 18 years of age or older.
* Signed informed consent form, which meets all criteria of current FDA regulations.
* If female and of child-bearing potential, have a negative urine pregnancy test at baseline visit, and prepare to abstain from sexual intercourse or use a reliable method of contraception during the study.
* A total score of at least 4 for the clinical signs and symptoms of tinea pedis for the target lesion. In addition, the most infected area must have a minimum score of at least 2 for erythema and a minimum score of at least 2 for scaling.
* A confirmed clinical diagnosis of tinea pedis with lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot.
* The presence of tinea pedis infection, confirmed by the observation of segmented fungal hyphae during a microscopic 10% potassium hydroxide wet mount examination.

Exclusion Criteria:

* Females who are pregnant, lactating or likely to become pregnant during the study.
* Use of antipruritics, including antihistamines within 72 hours prior to baseline visit.
* Use of topical corticosteroids, antibiotics or antifungal therapies within 2 weeks prior to baseline visit.
* Use of systemic corticosteroids, antibiotics or antifungal therapies within 1 month prior to baseline visit.
* Use of oral terbinafine or itraconazole within 2 months prior to baseline visit.
* Use of immunosuppressive medication or radiation therapy within 3 months prior to baseline visit.
* Any known hypersensitivity to Naftifine HCl, any component of the formulation or other antifungal agents.
* Confluent, diffuse moccasin-type tinea pedis of the entire plantar surface.
* Significant history or current evidence of chronic infectious disease, system disorder, organ disorder, or other medical condition that would place the patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
* Evidence of any concurrent dermatophytic infection of the toe nails or dermatological condition of the foot that may interfere with the evaluation of tinea pedis.
* Patients with a past history of tinea pedis infections with a lack of response to antifungal therapy.
* Patients who would be non-compliant with the requirements of the study protocol.
* Participation in a research study within 30 days prior to baseline visit.
* Employees or family members of employees of the research center or investigator.
* Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Therapeutic Cure | 42 Days
  Patients with both mycological cure and clinical cure at the final follow-up visit two weeks fter the end of treatment (Day 42) will be considered therapeutic cures.